CLINICAL TRIAL: NCT01484002
Title: Collaborative Analysis of UHMWPE Explants: Conventional UHMWPE With No Radiation and Marathon
Brief Title: Analysis of Crosslinked and Conventional Polyethylene Explants
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: Orthopaedic Biomechanics and Biomaterials Laboratory at Massachusetts General Hospital (Unknown); DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: AORI2011-0101; MGH Agreement No: A208947 (Other Grant/Funding Number: DePuy Orthopaedics, Inc.)
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis
Keywords: Hip replacement; Crosslinked and conventional polyethylene; Oxidation; Crosslink density; Outcome
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crosslinked polyethylene liners: Polyethylene liners from joint replacements that were crosslinked and heat treated to eliminate free radicals.
  Interventions: Device: Total hip arthroplasty
- Conventional polyethylene liners: Polyethylene liners from joint replacements that manufactured from conventional UHMWPE and terminally sterilized by methods that did not involve gamma-irradiation.
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Replacement of a patient's native hip with an artificial implant featuring a metal-on-polyethylene articulation
  Other Names: DePuy Marathon crosslinked polyethylene; DePuy Enduron conventional polyethylene

SUMMARY:
This retrospective study will investigate the changes that occur in ultrahigh molecular weight polyethylene (UHMWPE) implants that have been retrieved from joint replacement patients. Analysis techniques will include Fourier Transform Infrared Spectroscopy (FTIR), Differential Scanning Calorimeter (DSC) and crosslink density measurements. Crosslink density measurements will be evaluated as a function of distance away from the articular surface and the rim of the implant. Gel and hydroperoxide contents will also be evaluated. The objective is to characterize the in vivo and ex vivo changes that occur with cross-linked and conventional polyethylene bearings sterilized by methods that do not involve radiation. The investigators hypothesize that polyethylene absorbs lipids in vivo but experiences negligible oxidation or reductions in polymer crosslinking until it is explanted and stored at room temperature with access to ambient air.

DETAILED DESCRIPTION:
For many years, gamma-irradiation in air was a common method for the terminal sterilization of ultrahigh molecular weight polyethylene (UHMWPE) materials used for joint replacement. A serendipitous byproduct of sterilization with gamma-irradiation was polymer crosslinking that tended to improve the wear performance of the polyethylene. During the 1990s, however, the orthopaedic community became aware that gamma-irradiation created free radicals within polyethylene, rendering the material susceptible to oxidative degradation. In view of this potentially deleterious effect, terminal sterilization methods using chemical surface treatments were developed to avoid free radical formation. To induce polyethylene crosslinking without residual free radicals, manufacturers also developed methods to crosslink the polyethylene followed by heat treatments to eliminate free radicals. These crosslinked materials were introduce during the latter part of the 1990s and clinical outcome studies among hip replacement patients have demonstrated substantially reduced wear at early follow-up intervals based on radiographic measurements. However, the long-term performance of crosslinked polyethylene is unknown and some investigators have expressed concerns related to in vivo degradation. Additionally, some crosslinked UHMWPE components have shown high levels of oxidation and chain scission after removal from patients and storage in air. Among these implants, it is unknown whether the oxidation and chain scission occurred during implantation or after the polyethylene was removed from the patient.

This study will characterize the material properties of polyethylene liners retrieved from hip replacement patients. The study population will include crosslinked and conventional UHMWPE liners that were terminally sterilized without the use of radiation. To quantify the potential effects of different storage methods, liners that were vacuum packed and frozen after retrieval and others that were stored at room temperature with access to ambient light and air following explantation will be included in the study population. Analysis techniques will include Fourier Transform Infrared Spectroscopy (FTIR), Differential Scanning Calorimeter (DSC) and crosslink density measurements. Crosslink density measurements will be evaluated as a function of distance away from the articular surface and the rim of the implant. Gel and hydroperoxide contents will also be evaluated. The goal of the analysis is to better understand the changes in polyethylene material properties that occur in vivo and ex vivo.

ELIGIBILITY:
Inclusion Criteria:

* Retrieved total hip arthroplasty liners maintained by the Anderson Orthopaedic Research Institute
* Crosslinked or conventional liners terminally sterilized without gamma-irradiation

Exclusion Criteria:

* Liners terminally sterilized with gamma-irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crosslinked and conventional polyethylene liners terminally sterilized without gamma-irradiation will be used for this study. Specimens will be selected from the implant retrieval collection maintained by the Anderson Orthopaedic Research Institute.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oxidation levels | At an average of 5 years in vivo
  Polyethylene oxidation levels will be quantified as a function of depth away from the articular and rim surfaces using Fourier Transform Infrared Spectroscopy (FTIR). Pre and post-hexane and nitric oxide (NO) exposed post-hexane thin sections will be analyzed.

SECONDARY OUTCOMES:
Absorbed lipids | At an average of 5 years in vivo
  Absorbed lipids will be evaluated by determining the level of carbonyls before and after hexane extraction using Fourier Transform Infrared Spectroscopy (FTIR).
Crosslink density | At an average of 5 years in vivo
  Crosslink density will be evaluated using the gravimetric method on thin sections (~300μm) cut co-planar to the articular surfaces.
Differential Scanning Calorimeter (DSC) | At an average of 5 years in vivo
  Differential Scanning Calorimeter (DSC) will be used to determine the 1st and 2nd heats, and 1st cool crystallinity, peak melting/crystallization points.
Hydroperoxides | At an average of 5 years in vivo
  Hydroperoxides will be evaluated with FTIR by NO treatment after hexane extraction.
Vinyl end-groups | At an average of 5 years in vivo
  Vinyl end-groups will be evaluated with FTIR after hexane extraction to quantify chain scission.
Trans vinylene (TVI) unsaturations | At an average of 5 years in vivo
  Trans vinylene (TVI) unsaturations will be evaluated with FTIR after hexane extraction to determine radiation history and dose.
Crystallinity | At an average of 5 years in vivo
  Infra-red crystallinity will be evaluated with FTIR after hexane extraction.
Gel content | At an average of 5 years in vivo
  To quantify the extent of chain scission, gel content will be evaluated by measuring the non-extractable portion of the molecules using thin sections cut co-planar to the articular surfaces with a microtome and extracting the polyethylene chains from these sections in hot xylene.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hopper, Jr., PhD, Study Director — Anderson Orthopaedic Research Institute
Locations (2):
- United States (2):
  - Orthopaedic Biomechanics and Biomaterials Laboratory at Massachusetts General Hospital, Boston, Massachusetts
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia

REFERENCES:
- [Background] Muratoglu OK, Wannomae KK, Rowell SL, Micheli BR, Malchau H. Ex vivo stability loss of irradiated and melted ultra-high molecular weight polyethylene. J Bone Joint Surg Am. 2010 Dec 1;92(17):2809-16. doi: 10.2106/JBJS.I.01017. PMID 21123611
- [Background] Bargmann LS, Bargmann BC, Collier JP, Currier BH, Mayor MB. Current sterilization and packaging methods for polyethylene. Clin Orthop Relat Res. 1999 Dec;(369):49-58. doi: 10.1097/00003086-199912000-00006. PMID 10611860
- [Background] Currier BH, Van Citters DW, Currier JH, Collier JP. In vivo oxidation in remelted highly cross-linked retrievals. J Bone Joint Surg Am. 2010 Oct 20;92(14):2409-18. doi: 10.2106/JBJS.I.01006. PMID 20962191
- [Background] Currier BH, Currier JH, Mayor MB, Lyford KA, Collier JP, Van Citters DW. Evaluation of oxidation and fatigue damage of retrieved crossfire polyethylene acetabular cups. J Bone Joint Surg Am. 2007 Sep;89(9):2023-9. doi: 10.2106/JBJS.F.00336. PMID 17768201
- [Background] Engh CA Jr, Stepniewski AS, Ginn SD, Beykirch SE, Sychterz-Terefenko CJ, Hopper RH Jr, Engh CA. A randomized prospective evaluation of outcomes after total hip arthroplasty using cross-linked marathon and non-cross-linked Enduron polyethylene liners. J Arthroplasty. 2006 Sep;21(6 Suppl 2):17-25. doi: 10.1016/j.arth.2006.05.002. PMID 16950057
- [Background] Malchau H, Bragdon CR, Muratoglu OK. The stepwise introduction of innovation into orthopedic surgery: the next level of dilemmas. J Arthroplasty. 2011 Sep;26(6):825-31. doi: 10.1016/j.arth.2010.08.007. Epub 2010 Oct 2. PMID 20888183
- See also: Website for the Anderson Orthopaedic Research Institute — http://aori.org